CLINICAL TRIAL: NCT01613352
Title: Same Day Discharge After Surgery for Early Breast Cancer - a Feasible Option
Brief Title: Feasibility of Ambulatory Surgery for Early Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Jaana Vironen, Associate chief surgeon, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 329 / E6 / 07
Record Dates: First submitted 2012-06-05; First posted 2012-06-07 (Estimated); Last update posted 2012-06-07 (Estimated); Status verified 2012-06

CONDITIONS: Early Breast Cancer; Psychosocial Wellbeing; Ambulatory Surgery
Keywords: Early breast cancer surgery; Psychosocial wellbeing; Ambulatory surgery
MeSH Terms: conditions — Breast Neoplasms | interventions — Ambulatory Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Day surgery group (Experimental): Patients who underwent breast conserving surgery and sentinel node biopsy only and were randomized to ambulatory surgery group.
  Interventions: Other: Ambulatory surgery
- In-Patient group (Active Comparator): Patients who underwent breast conserving surgery and sentinel node biopsy only and were randomized to in-patient group.
  Interventions: Other: Ambulatory surgery

INTERVENTIONS:
Other: Ambulatory surgery — Sentinel node mapping was done on the previous day and the patients were operated on first in the morning.

SUMMARY:
The aim was to assess the patient compliance and medical and psychosocial effects of same day hospital discharge after breast conserving surgery and sentinel node biopsy only.

DETAILED DESCRIPTION:
The patients with small breast tumours (<2 cm)and clinically node negative disease, were randomized to receive breast conserving surgery and sentinel node biopsy as ambulatory surgery or inpatient-surgery.Complication rate, patient satisfaction and psychosocial outcomes were compared. The psychosocial effects of the treatment mode on their spouses were recorded as well.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer < 2cm
* Clinically node negative
* ASA I-II

Exclusion Criteria:

* Axillary clearance performed
* ASA III-IV
* No adult companion at home

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-03; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Psychosocial wellfare | First postoperative day
  Difference between the groups in questionnaire measuring anxiety and psychosocial wellfare

SECONDARY OUTCOMES:
Number of complications and return to hospital rate | one week
  The difference in the number of complications or return to the hospital rate between the groups

CONTACTS AND LOCATIONS:
Overall Officials: Jaana H Vironen, MD, PhD, Principal Investigator — Helsinki University Central Hospital, Jorvi Hospital
Locations (1):
- Helsinki University Central Hospital, Jorvi Hospital, Espoo, HUS, Finland

REFERENCES:
- [Derived] Ojala K, Vironen JH, Mattila K, Eklund AM, Leidenius MH, Meretoja TJ. Feasibility of Day Surgery in Patients With Breast Conservation and Sentinel Node Biopsy: A Randomized Controlled Trial. Scand J Surg. 2016 Mar;105(1):29-34. doi: 10.1177/1457496915583201. Epub 2015 Apr 28. PMID 25922474